CLINICAL TRIAL: NCT02983643
Title: Body Composition Changes During Stem Cell Transplantation: The Case Of Lymphoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Aix Marseille Université (Other)
Responsible Party: Sponsor
Other Study IDs: IM.J-EC.04
Record Dates: First submitted 2016-10-03; First posted 2016-12-06 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2016-10

CONDITIONS: Hematopoietic Stem Cell Transplantation; Malnutrition; Metabolic Syndrome
Keywords: Skeletal Muscle Index; Visceral Adipose Tissue; Metabolic Syndrome
MeSH Terms: conditions — Malnutrition; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Skeletal Muscle Index (SMI) and Visceral Adipose Ratio (VAR) assess body composition changes and disclose malnutrition risk effectively. The aims of the study are to assess prevalence of malnutrition in patients planned for SCT, to characterize changes in body composition (SMI, total adipose tissue and VAR) that occur in the peri transplantation phase, and to identify Waist Circumference (WC) cut off points associated with the metabolic syndrome (MetSyn) in patients with B and T cell Lymphoma.

DETAILED DESCRIPTION:
This study is a retrospective cohort study of patients having B and T cell lymphoma, who underwent SCT in the Bone Marrow Transplantation (BMT) unit at AUBMC. Consecutive patients having B and T lymphoma who underwent SCT at AUBMC will be identified by the research team and will be included as per the below inclusion and exclusion criteria. Starting from June 2016, patients who meet the inclusion criteria will be included in the study up until June 2006.

The radiologist will access the AUBMC PACS system to review PET/CT scans of the identified patients. SMI, visceral, subcutaneous and intramuscular adipose tissues will be established by assessing at the level of L3.

ELIGIBILITY:
Inclusion Criteria:

* Age>16 years
* Patients having B and T cell lymphoma who have undergone SCT at AUBMC

Exclusion Criteria:

* Patients with a missing pre-SCT PET/ CT scan
* Patients with 2 missing post SCT PET / CT scan

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients having B and T lymphoma who underwent SCT between January 2006 and June 2016 at AUBMC are identified by the research team and are included as per the below inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Sarcopenia Prevalence | 3 months post Stem Cell Transplantation
Skeletal Muscle Index Changes | 3 months post Stem Cell Transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Jean El Cheikh, MD, Principal Investigator — AUBMC
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes